CLINICAL TRIAL: NCT01850927
Title: Effect of Remote Ischemic Preconditioning on Subclinical Myocardial Injury in Major Abdominal Surgery: a Randomised Controlled Trial
Brief Title: Perioperative Reduction of Inapparent Myocardial Injury
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Surgical Research Group (Other)
Collaborators: Royal Berkshire NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSRG-002
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-03

CONDITIONS: Perioperative Myocardial Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Patients will receive remote ischaemic preconditioning prior to surgery. After the induction of anaesthesia, a blood pressure cuff will be placed on an upper arm and inflated to 200mmHg for 5 minutes, then deflated for 5 minutes, repeated for a total of 3 inflation-deflation cycles.
  Interventions: Procedure: Remote ischaemic preconditioning
- Control (Sham Comparator): Patients will have the same procedure as for the intervention group, however the blood pressure cuff valve will be left open throughout the 30 minute treatment. Patients will be kept under anaesthesia for this additional time.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning
  Arms: Intervention
Procedure: Control
  Arms: Control

SUMMARY:
Recent data suggests that subclinical myocardial injury occurs in patients undergoing major abdominal surgery, and the degree of damage is proportionally linked to morbidity and mortality in the short and medium terms. Therefore, new methods of limiting myocardial damage are urgently needed.

Ischemic preconditioning is a phenomenon whereby a brief non-lethal ischemia-reperfusion stimulus gives a protective effect to further ischemic insults. In remote ischemic preconditioning (RIPC), this initial stimulus is carried out away from the region of interest, normally a limb. In meta-analysed syntheses the effect size of RIPC in reducing cardiac damage during bypass grafting, as characterised by troponin release, seems to be about 35%.

The PRIME Study will assess the value of RIPC in reducing subclinical myocardial injury in patients undergoing major abdominal surgery. Post-operative troponin release will be used as a surrogate marker of myocardial damage. There is no good data on which to build a reliable sample size calculation, therefore we estimated samples sizes using supplementary data from the recent VISION study. The investigators intend to build a clinically powered study from the results of this study.

Study design will be by single-centre single-blind randomised control trial. Allocation will be 1:1. All treatments will be carried after induction of anaesthesia, prior to surgery. In the RIPC-treatment group, a blood pressure cuff inflated on an upper limb to 200mmHg for 5 minutes, and then deflated for 5 minutes, repeated in three cycles. In the control group, the blood pressure cuff will not be inflated, but the patient will remain under anaesthesia for the same amount of time.

Primary endpoint will be peak post-operative 5th generation hs-TnT (highly sensitive Troponin-T, ng/ml). Secondary endpoint will be hs-TnT area-under-the-curve, major adverse cardiovascular events, serious surgical complications, non-cardiovascular death, quality of life, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* is ≥ 45 years old;
* is undergoing elective major colorectal or upper GI surgery.

Exclusion Criteria

* Diabetic patients that are taking glibenclamide medication
* Patients with upper limb peripheral vascular disease, including those with arteriovenous fistula for dialysis
* Untreated hypertension (defined as two or more readings >180mmHg systolic on admission for surgery)
* Current participation in any study investigating troponin levels or ischaemic preconditioning
* Unable or lacks capacity to give informed consent to participation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Peak post-operative troponin (ng/L) | At 6-12, 24, 48, 72h

SECONDARY OUTCOMES:
Any major adverse cardiovascular events | 30 days
  "MACCE" - defined as any new arrhythmia, myocardial infarction, congestive heart failure, angina, stroke or non-fatal cardiac arrest, or cerebrovascular or cardiovascular death
Any serious surgical complications | 30 days
  'SSG' - defined as any post-operative complication requiring radiological, surgical, or endoscopic intervention, or intensive care, or leading to non-vascular death (i.e. Calvien-Dindo III-V).
Area-under-the-curve post-operative troponin (ng/L) | 72 hours
Positive post-operative troponin (binary endpoint, >20ng/L) | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Walden, MBBS PhD MRCP, Study Director — Royal Berkshire Hospitals; Stefan S Antonowicz, MBChB MRCS, Principal Investigator — Royal berkshire Hospitals
Locations (1):
- Royal Berkshire Hospital, Reading, Berks, United Kingdom

REFERENCES:
- [Derived] Antonowicz SS, Cavallaro D, Jacques N, Brown A, Wiggins T, Haddow JB, Kapila A, Coull D, Walden A. Remote ischemic preconditioning for cardioprotection in elective inpatient abdominal surgery - a randomized controlled trial. BMC Anesthesiol. 2018 Jun 26;18(1):76. doi: 10.1186/s12871-018-0524-6. PMID 29945555